CLINICAL TRIAL: NCT01101555
Title: A Randomised, Single-blind, Placebo-controlled, Study Toevaluate the Safety, Tolerability, Pharmacodynamics Andpharmacokinetics of Repeat Subcutaneous Administration Ofotelixizumab in Subjects With Rheumatoid Arthritis
Brief Title: Repeat Dose Subcutaneous Rhumatoid Arthritis Efficacy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 113299
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid arthritis; repeat dose; pharmacodynamics; pharmacokinetics; subcutaneous; safety; Otelixizumab; long term follow up; tolerability
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- COHORT 1: CUMULATIVE DOSE 1.5MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 3 days, dose 0.3, 0.5, 0.7, four patients in cohort, one of which is on placebo, escalation increment N/A
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 2: CUMULATIVE DOSE 3.5MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 5 days, dose 0.3, 0.5, 0.7, 1.0, 1.0 four patients in cohort, one of which is on placebo, escalation increment 2.3 fold.
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 3: CUMULATIVE DOSE 6.0MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 7 days, dose 0.3, 0.7, 5 x 1.0 four patients in cohort, one of which is on placebo, escalation increment 1.7 fold.
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 4: CUMULATIVE DOSE 8.0MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 5 days, dose 0.3, 0.7, 1.0, 2 x 3.0 four patients in cohort, one of which is on placebo, escalation increment 1.33 fold.
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 5: CUMULATIVE DOSE 10MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 10 days, dose 10 x 1.0 four patients in cohort, one of which is on placebo, escalation increment 1.25 fold.
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 6: CUMULATIVE DOSE 15MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 15 days, dose 15 x 1.0 six patients in cohort, one of which is on placebo, escalation increment 1.5 fold.
  Interventions: Drug: subcutanious administration; Other: Placebo
- COHORT 7: CUMULATIVE DOSE 15MG, ADMINISTERED SUBCUTANEOUSLY (Experimental): Duration of treatment 5 days, dose 5 x 3.0 six patients in cohort, one of which is on placebo, escalation increment N/A
  Interventions: Drug: subcutanious administration; Other: Placebo

INTERVENTIONS:
Drug: subcutanious administration — drug will be administered subcutaneously in varying amounts over a verying time period according to details stated in the 'arms' section
Other: Placebo — Placebo will be given to one member of each cohort.

SUMMARY:
This study is a randomised, single-blind, placebo-controlled, repeat dose study of otelixizumab administered subcutaneously in rheumatoid arthritis patients. One cohort will receive a single dose of adalimumab (HUMIRA, Abbott) as rescue medication to assess additional concomitant safety and tolerability issues.

DETAILED DESCRIPTION:
Otelixizumab is a humanized, aglycosyl, non-mitogenic, anti CD3 monoclonal antibody (MAb) directed against the ε domain of the human lymphocyte antigen CD3, which is currently undergoing phase III clinical trials in adult new-onset type I diabetes mellitus patients and has been evaluated in rheumatoid arthritis and psoriasis patients in small exploratory studies. Otelixizumab has been administered via the subcutaneous route as a single dose in type I diabetes patients. This study is a randomised, single-blind, placebo-controlled, repeat dose study of otelixizumab administered subcutaneously in rheumatoid arthritis patients. One cohort will receive a single dose of adalimumab (HUMIRA, Abbott) as rescue medication to assess additional concomitant safety and tolerability issues.

This study will consist of a screening phase, followed by an in-house phase whereby otelixizumab will be administered to cohorts in a staggered fashion. Six cumulative doses will be evaluated covering a 10-fold dose range in seven cohorts. The starting regimen will be three doses (1.5 mg cumulative dose), increasing to 15 doses (15 mg cumulative dose). Cohorts 1a and 1b have been included as optional lower doses. Serial blood samples will be obtained for clinical laboratory testing, determination of pharmacodynamic markers, serum otelixizumab PK parameters, and immunogenicity. Safety and pharmacodynamic data from the previous dose(s) will be evaluated prior to dose escalation or modification to ensure safety and to achieve target systemic peripheral blood pharmacology. Adverse events, laboratory values, vital signs and ECG's will be monitored closely during this study. All subjects in the study will undergo long-term follow-up out to 48 months to monitor and ensure patient safety.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female subjects between 18 and 75 years of age inclusive.
2. A female subject is eligible to participate if she is of:

   1. Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 mIU/ml and estradiol <40 pg/ml (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   2. Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1.1 for an appropriate period of time to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception for at least two weeks prior to dosing and for at least 60 days after the last dose.
3. Male subjects must agree to use one of the contraception methods listed in Section 8.1.2. This criterion must be followed from the time of the first dose of study medication until at least 60 days after the last dose of otelixizumab or two months after adalimumab (Cohort 6 only).
4. Body mass index within the range 18.5 - 35 kg/m^2 inclusive
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form and willing and able to follow the procedures outlined in the protocol.
6. A 12-lead ECG at pre-study screening measured in triplicate, which in the opinion of the Principal Investigator or physician designee has no abnormalities that will compromise safety in this study. QTcB < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
7. No significant and/or active disease in any body system. Examples of significant diseases include but are not limited to: coronary artery disease, congestive heart failure, uncontrolled hypertension, emphysema, seizure disorder, chronic infectious disease ( e.g., chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis (TB) or latent tuberculosis, hepatitis B and C).
8. The subject has a diagnosis of RA according to the revised 1987 criteria of the American College of Rheumatology
9. The subject tests positive for Rheumatoid factor
10. The subject has not previously received otelixizumab or any other anti-CD3 monoclonal antibody, e.g., OKT3 (muromonab or Orthoclone), ChAglyCD3, or hOKT3γ1 (ala ala), and is willing to refrain from using any such antibody for 2 years after the last dose of study drug unless invited to participate in possible future studies with otelixizumab.
11. If taking methotrexate, the patient must have been taking methotrexate for at least 12 weeks and to be on a stable dose of methotrexate (7.5-25 mg/week) for at least four weeks prior to dosing and be willing to remain on this dose until day 28 of the study unless change required for clinical management of disease activity or safety.
12. If sulfasalazine is being taken, the patient must have been taking sulfasalazine for at least 12 weeks and to be on a stable dose within local treatment guidelines for at least four weeks prior to dosing and be willing to remain on this dose until day 28 of the study unless change required for clinical management of disease activity or safety.
13. If leflunomide is being taken, the patient must have been receiving this DMARD for at least six months prior to dosing with otelixizumab and the DMARD dose has been stable dose within local treatment guidelines for four weeks prior to dosing with study drug and be willing to remain on this dose until day 28 of the study unless change required for clinical management of disease activity or safety.
14. Patients on glucocorticoids e.g. prednisolone (≤10mg/day), must be on stable dosing regimens for at least four weeks prior to dosing and be willing to remain on this dose until day 28 of the study.
15. PRN use is acceptable for NSAIDS and COX-2 inhibitors within local treatment guidelines. Chronic NSAID/COX-2 inhibitor use is not permitted.
16. The subject is seropositive for EBV with <10,000 copies of EBV DNA per 106 lymphocytes (qPCR) or seronegative with no evidence of recent EBV exposure (EBV IgM negative and no clinical symptoms suggestive of acute infection)
17. The subject has no current or prior malignancy, other than non-melanoma skin cancer (subject must have had fewer than 5 occurrences of non-melanoma skin cancer, and the last occurrence must not be within 3 months of study entry).

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subjects with a history of significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, or Felty's syndrome)
2. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening; current or chronic history of liver disease.
3. The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
4. A positive test for HIV antibody or risk factors which predispose subject to HIV infection.
5. A positive test for syphilis according to local guidelines.
6. History of regular alcohol consumption within 6 months of the study defined as:

   • an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) or planning to take any investigational drug within six months of the last dose of study drug
8. The subject is currently receiving or has received an anti-rheumatic biological therapy within the following specified periods prior to dosing:

   Within four weeks:
   * Glucocorticoid unless given in doses equivalent to <=10 mg of prednisolone/day
   * Intramuscular. or i.v. corticosteroids
   * Live/attenuated vaccinations
   * Cyclosporine
   * Etanercept
   * Anakinra

   Within eight weeks:
   * Infliximab
   * Rituximab
   * Abatacept
9. Previous or current exposure to biologic cell-depleting anti-rheumatic therapies, including investigational compounds (e.g. anti-CD11a, anti-CD-20, anti-CD22, anti-BLyS/BAFF, anti-CD3, anti-CD5, anti-CD52).
10. Previous or current exposure to adalimumab.
11. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
12. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
13. Where participation in the study would result in donation of blood or blood products in excess of 600 mL within a 56 day period.
14. Pregnant females as determined by positive (serum or urine) hCG test at screening or prior to dosing, or lactating females.
15. The subject has received immunization with a vaccine within four weeks before the first dose of study medication or requires a vaccine within 30 days after the last dose of study medication.
16. A CD4+ lymphocyte count outside the range of (0.53 - 1.76 × 10^9 )/L during Screening.
17. The subject has had a significant systemic infection during the 6 weeks before the first dose of study drug (e.g., infection requiring hospitalization, major surgery, or IV antibiotics to resolve); other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-by-case basis by the investigator regarding whether they are serious enough to warrant exclusion).
18. The subject has received a course of oral antibiotics within 2 weeks of dosing day one.
19. History of recurrent or chronic infection.
20. The subject has had a splenectomy.
21. Subjects with a screening chest X-ray suggestive of TB without documentation of adequate TB treatment will be excluded.

    Screening for latent TB infection using intradermal injection of tuberculin (e.g. the Mantoux test or equivalent) should be conducted in accordance with local guidelines. The tuberculin skin test results should be evaluated according to the criteria for immunocompromised subjects. Subjects with a positive skin tuberculin test should be excluded if the investigator judges the patient to be at risk of latent TB infection). Cohort 6 are required to undergo radiographic screening with CXR, this is optional according to local guidelines for all other cohorts.
22. The subject has undergone any major surgical procedure within the 8 weeks before signing the consent form, or planning to undergo any such surgery within the 3 months after the last dose of study drug.
23. Positive plasma / white cell JC virus (JCV) PCR (either compartment)
24. The subject has a condition or situation that, in the investigator's judgment, is likely to cause the subject to be unable or unwilling to participate in study procedures or to complete all scheduled assessments.
25. Predisposition to thromboembolic disease, or thromboembolic event (excluding superficial) in past 12 months.
26. Has clinically significant cardiovascular and/or cerebrovascular disease, including but not limited to:

    * Previous history of stroke or transient ischaemic attack
    * Active unstable coronary artery disease within the last 6 months
    * Documented myocardial infarction in the 1 year prior to screening
    * Any cardiac surgery including percutaneous transluminal coronary angioplasty, coronary

    artery bypass grafting within a year prior to screening
    * Unstable angina
    * Clinically significant arrhythmia or valvular heart disease within previous year
    * Congestive heart failure with New York Heart Association Class II to IV symptoms. Class I is acceptable.
    * Untreated hypertension with systolic pressure greater than 160mmHg, and/or diastolic pressure greater than 95 mmHg.
27. The subject has clinically significant abnormal laboratory values during the Screening period, other than those due to RA. Abnormal values are permitted if, upon re-test, the abnormality was resolved
28. Liver Function Tests must not be outside the range: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin ≤ 1.5x ULN (isolated bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-05-12 (Actual); Primary Completion 2011-09-16 (Actual); Study Completion 2012-11-29 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 1 month
Change from baseline and number of subjects outside the normal range for blood pressure, heart rate, temperature, electrocardiography parameters (12-lead) | 1 month
Change from baseline in clinical chemistry and haematology parameters | 1 month
Epstein-Barr Virus viral load | 1 month
Individual absolute and percentage circulating peripheral T lymphocytes and CD4+ and CD8+ subset counts | 1 month
Saturation of CD3 antigen on peripheral blood T cells | 1 month

SECONDARY OUTCOMES:
Individual serum concentrations of otelixizumab and data permitting summary PK parameters | 1 month
Serum levels of anti-otelixizumab binding antibodies. Where binding antibodies are detected, proportion which are anti-otelixizumab neutralising antibodies. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113299 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/113299?search=study&search_terms=113299#rs
- Available data/document: Clinical Study Report: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113299 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register